CLINICAL TRIAL: NCT06886867
Title: Physical Function in Older Adults: Exergaming vs. Usual Care in Physical Therapy - A Randomized Controlled Trial
Brief Title: Comparing Exergaming and Usual Care Physical Therapy in Nursing Home Residents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBA-02
Record Dates: First submitted 2025-03-03; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Older Adults Institutionalized in Residential Homes
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): This group will perform approximately 28 minutes of exergaming 3 times a week for 6 weeks
  Interventions: Other: Exergaming
- Usual physical therapy care (Active Comparator): This group will perform their usual care exercises treatments for approximately 28 minutes for 3 times a week for 6 weeks
  Interventions: Other: Usual physical therapy care

INTERVENTIONS:
Other: Exergaming — Exergaming: Participants will perform different exercises through videogames
  Arms: Exergaming
Other: Usual physical therapy care — Usual care: Different exercises will be performed
  Arms: Usual physical therapy care

SUMMARY:
The objective of this clinical trial is to compare the effects of exergaming and usual care physical therapy on physical function in older adults residing in nursing homes.

This trial seeks to answer the following key questions:

* Does physical function differ between interventions after treatment?
* How do these interventions impact enjoyment of therapy?
* Are there differences in adherence or perceived exertion between the interventions?

DETAILED DESCRIPTION:
A single-blind, randomized controlled trial will be conducted to compare exergaming and usual care interventions. Participants will be recruited from nursing homes in the province of Toledo, and the study will follow the CONSORT guidelines for clinical, crossover, and parallel trials.

Two experimental groups will be tested, with interventions performed three days per week for six weeks, each session lasting approximately 30 minutes. The exergaming group will play seven video games from the Party Fowl app, while the usual care group will continue their standard exercise routine.

Outcome measures will be assessed at baseline, post-intervention (6 weeks), and at a 3-month follow-up to evaluate the middle-term effects of both interventions.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 60 years of age
* score equal to or greater than 20 on the Mini Mental cognitive test
* Subjects that present the ability to stand without the use of technical aids or with the technical assistance of a device used for walking.

Exclusion Criteria:

* severe visual impairment
* medical contraindication for physical activity
* pathology or problem that could prevent the test from being carried out.

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Physical function | Baseline, post-intervention (6 weeks) and 3 months follow-up.
  Physical function will be assessed using the Short Physical Performance Battery (SPPB)

SECONDARY OUTCOMES:
Hand grip strength | Baseline, post-intervention (6 weeks) and 3 months follow-up.
  Hand grip strength will be assessed using a hand dynamometer.
Exercise enjoyment | Post-intervention (6 weeks)
  This outcome will be measured Physical Activity Enjoyment Scale (PACES). Higher values indicate higher perceived satisfaction/ enjoyment.
Rate of Perceived Exertion | RPE will be measured inmediatley after the intervention
  Rate of perceived exertion will be measured using Borg (RPE 1-10). Higher values indicate higher levels of perceived exertion
Adherence | Through study completion (6 weeks), with a final adherence percentage calculated at the end of the intervention.
  Adherence will be measured by the percentage of sessions attended of each participant.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Nueva Esperanza Nursing Home, Fuensalida, Toledo
  - Universidad de Castilla-La Mancha, Toledo

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided to other researchers if asked to the principal investigator